CLINICAL TRIAL: NCT01482546
Title: Randomized Cross-Over Comparing Clinical Performance of Novice Trainee Endoscopists Using Conventional Air Insufflation Versus Warm Water Infusion Colonoscopy
Brief Title: Comparing Clinical Performance of Novice Trainee Endoscopists Using Conventional Air Insufflation Versus Warm Water Infusion Colonoscopy
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 238499
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Colonoscopy Education
Keywords: colonoscopy; trainees; water; adenoma detection rate; cecal intubation rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Water Colonoscopy Method: As first described by Dr. Felix W. Leung, the maneuvers can be summarized as warm water infusion in lieu of air insufflation combined with suction removal of all residual colonic air and residual feces by water exchange. The air pump will be turned off before insertion of the colonoscope into the rectum to avoid accidental insufflation of air. Warm water (at 36-37ºC) maintained using a water bath and heat saver envelop will be infused intermittently. The minimum amount of water needed to distend the colon and open the lumen will be used during scope insertion. Cecal intubation will be suggested by appropriate movement of the endoscopic image on the monitor screen when the right lower quadrant is palpated or the appendiceal orifice visualized under water. The cecum will then be distended by air to confirm visualization of the ileocecal valve and appendiceal orifice. No specific limit will be set for the volume of water to be used.
- Air Colonoscopy Method: The minimal amount of air will be used during insertion to open the lumen. Minimal amounts of water (10 to 50 mL) at room temperature will be used for washing of residual feces. If insertion is hindered by scope looping, attempts at loop reduction will be made. If advancement does not occur within 3 to 5 minutes, an assistant will provide abdominal compression, followed by changing the patient's position to facilitate passage of the colonoscope. Cecal intubation will be suggested by identification of the appendiceal orifice and ileocecal valve or intubation of the terminal ileum.

SUMMARY:
Hypothesis: Novice trainees will achieve significantly higher clinical competence and patient satisfaction scores with the use of warm water infusion method when compared with traditional air insufflation

Primary outcome: adenoma detection rate

Secondary outcomes: (1) independent cecal intubation rate, (2) trainer assessment of trainee's colonoscopy skills, (3) trainee's assessment of clinical confidence, (4) procedural medication requirement, (5) patient pain level during procedure, (6) patient satisfaction at procedure completion, and (7) patient willingness to repeat procedure'

Specific Aim: To demonstrate the stated hypothesis via above outcome measures. The long term goal is to provide evidence to influence other training institutions to consider education in the warm water infusion method'

DETAILED DESCRIPTION:
Study Design: Prospective randomized cross-over study in a university based setting (University of California Davis, Sacramento, California) with a diverse patient population.

Participants: Total of 6 first year gastroenterology trainees (3 enrollees per year from July 2011 to July 2012)

Recruitment: Trainees' names and contact information will be acquired via the program director. They will be contacted in person on the first day of their fellowship orientation and provided information regarding the study.

Randomization: A sealed envelope containing the randomized method (conventional air insufflation or warm water infusion) will be opened at the time of signed consent for study participation.

Cross-over Design: Trainees will perform colonoscopies using the randomized method with a dedicated attending physician who uses air and/or water method as part of standard clinical practice for 6 months, at which point they will cross-over to the alternate method of colonoscopy with another dedicated attending for the remaining 6 months of their first year of fellowship.

Air Insufflation Method:

The minimal amount of air will be used during insertion to open the lumen. Minimal amounts of water (10 to 50 mL) at room temperature will be used for washing of residual feces. If insertion is hindered by scope looping, attempts at loop reduction will be made. If advancement does not occur within 3 to 5 minutes, an assistant will provide abdominal compression, followed by changing the patient's position to facilitate passage of the colonoscope. Cecal intubation will be suggested by identification of the appendiceal orifice and ileocecal valve or intubation of the terminal ileum.

Warm Water Infusion Method:

As first described by Dr. Felix W. Leung, the maneuvers can be summarized as warm water infusion in lieu of air insufflation combined with suction removal of all residual colonic air and residual feces by water exchange. Because insufflated air could lengthen the colon and exaggerate angulations at the flexures making insertion more difficult, the air pump will be turned off before insertion of the colonoscope into the rectum to avoid accidental insufflation of air. Further minimization of angulations at the flexures can be achieved by suction removal of all encountered residual air. Warm water (at 36-37ºC) maintained using a water bath and heat saver envelop will be infused intermittently using an Olympus OFP peristaltic flushing pump via an EndoGator auxiliary water port connector and disposable water bottle system for Olympus scopes. The minimum amount of water needed to distend the colon and open the lumen will be used during scope insertion. When the luminal water becomes turbid due to residual feces, the discolored water will be suctioned and replaced by clean water until the lumen is visualized again. If advancement does not occur within 3 to 5 minutes, an assistant will provide abdominal compression, followed by changing the patient's position to facilitate passage of the colonoscope. Cecal intubation will be suggested by appropriate movement of the endoscopic image on the monitor screen when the right lower quadrant is palpated or the appendiceal orifice is visualized under water. The cecum will then be distended by air to confirm visualization of the ileocecal valve and appendiceal orifice. No specific limit will be set for the volume of water to be used.

Colonoscopy Procedures:

Trainees randomized to either use of conventional air insufflation or warm water infusion method will be performing colonoscopies with a dedicated endoscopy attending during their half-day weekly outpatient endoscopy clinics (for which main indications for colonoscopy will be screening or surveillance) for each 6-month study period. Three faculty gastroenterologists will be participating as dedicated research personnel.

Patients will be monitored in a standard fashion (including regular nursing assessments of vital signs and discomfort). The sedation nurse will administer medications during the procedure according to patient pain levels (0=none to 10=most severe) assessed every 3-5 minute intervals or at any time the patient appears to be in discomfort. Standard incremental doses of medications (using either meperidine 25mg or fentanyl 25 mcg and midazolam 1mg) will be offered to the patient when the pain level is ≥ 2. The nurse will record procedural times (start time, cecal intubation time, and end time in minutes), medications administered (for pre-procedural sedation, from procedure start to cecal intubation, and during withdrawal period from cecum to across anus), and attending involvement (hands-on assistance or take-over).

An attending dedicated to colonoscopy training will be present for the entire duration of the procedure. Cecum is considered reached by the attending if clear-cut cecal landmarks are identified (appendiceal orifice, ileocecal valve, or intubation of the terminal ileum). In concordance with prior studies, attending endoscopists will allow trainees 20 minutes to reach the cecum, provided the examination is progressing in a safe manner and the patient is comfortable. If advancement does not occur within 3 to 5 minutes, an assistant will provide abdominal compression, followed by changing the patient's position to facilitate passage of the colonoscope. If the trainee has not reached the cecum by 20 minutes, the instructor will take over until the cecum is reached. The instructor will take over sooner than this if the trainee cannot advance the colonoscope for 5 minutes at the same site, or if it is judged that patient tolerance is becoming a factor. For both the air and water methods, unlimited verbal instruction will be allowed so that the instructor may guide the trainee with descriptions of maneuvers as if he/she were performing the procedure. The instructor will not provide hands-on assistance until either the trainee stated that he or she had reached the cecum, 20 minutes had passed, or it was necessary for the instructor to take over sooner than 20 minutes for one of the reasons stated above.

After each colonoscopy, the instructor will fill out a questionnaire regarding any prior colonic surgery, presence of abnormal anatomy or masses, polyp detection and removal, quality of preparation using the Boston Bowel Preparation Scale, and difficultly of the procedure (1=very easy to 5=very difficult). Overall assessment of the trainee's colonoscopy skills will be assessed by the instructor after each procedure (1=poor to 5=excellent). The instructor will also indicate whether the cecum was intubated and the colonoscopy completed independently by the trainee, if there was hands-on assistance, or if attending had to take-over the procedure. The trainee will be assessed for ease of learned technique (1=very easy to 5=very difficult) and self-assessment of clinical confidence (1=not at all confident to 5=extremely confident).

Record Keeping and Standardization:

A data collection sheet will be used for each study case, which includes data to be recorded by sedation nurse (procedural times, patient pain scores, medications administered, instructor involvement, and volume of water used), trainee self-evaluation, and attending evaluation of the case and trainee skill. A short post procedural survey that will be provided to patients to assess post-procedural pain, experience, satisfaction, and willingness to undergo repeat procedure. In addition to photographic images documenting cecal intubation that are scanned into our electronic records, a digital video recorder will be used to record all procedures so that the consultant and PI/investigators may review a predetermined 10% of the cases to ensure a uniform standard of reporting times, quality of preparation, polyp detection, and degree of difficulty. Personal identifiers will be removed from all digital images captured. We will track the number of additional colonoscopies that the trainee will perform as part of their inpatient rotations so that it may later be analyzed as a potential confounder. Pathology reports for all removed specimens will be recorded so that adenoma detection rates may be determined.

Statistical Analysis Plan:

Chi-squared (χ2) or Fisher's exact test analysis will be used to compared the proportion of successful trainee unassisted cecal intubation cases (primary outcome) between the conventional air insufflation and warm water infusion colonoscopy methods. Secondary outcome variables will be compared using Chi-squared test, Fisher's exact test or Mann Whitney U test as appropriate. Multivariate logistic regression analysis will be used to evaluate factors affecting cecal intubation time and success. We will also calculate the trainees' learning curves in consecutive blocks of 25 procedures (for air and water methods) using one-way variance analysis and Tukey Honestly Significant Difference test to compare unassisted cecal intubation and colonoscopy success rates and time required for cecal intubation and withdrawal as previously reported for conventional air method.

ELIGIBILITY:
Inclusion Criteria:

* Novice endoscopists without prior colonoscopy experience

Exclusion Criteria:

* Trainees who do not meet the basic prerequisites as stated above, or who are not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First Year Gastroenterology Trainees
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate | two years

SECONDARY OUTCOMES:
independent cecal intubation rate | two years

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States